CLINICAL TRIAL: NCT07061496
Title: Comparative Effects of Exercise and Metformin on Glycemic Control in Prediabetic Adults: A Community-Based, Open-Label, Randomized Trial in a Low-Resource Setting
Brief Title: Comparative Effects of Exercise and Metformin on Glycemic Control in Prediabetic Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umair Ali (Other Government)
Collaborators: CMH Nowshera (Unknown)
Responsible Party: Sponsor-Investigator, Umair Ali, Dr, Combined Military Hospital Nowshera
Organization: Combined Military Hospital Nowshera (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMHNSR-REF-17
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Pre Diabetic; Pre Diabetes
Keywords: Pre diabetic; Exercise; Metformin
MeSH Terms: conditions — Glucose Intolerance; Motor Activity | interventions — Metformin; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): Moderate aerobic activity (e.g., brisk walking) for 30-45 minutes/day, 5 days/week, for 12 weeks.
  Interventions: Behavioral: Moderately intense exercise
- Metformin Group (Active Comparator): Participants will receive oral metformin 500 mg twice daily for 12 weeks.
  Interventions: Drug: MetFORMIN 500 Mg Oral Tablet

INTERVENTIONS:
Behavioral: Moderately intense exercise — Structured moderate-intensity aerobic activity (e.g., brisk walking) for 30-45 minutes/day, 5 days/week, for 12 weeks.
  Other Names: Exercise Group
  Arms: Exercise Group
Drug: MetFORMIN 500 Mg Oral Tablet — Participants will receive oral metformin 500 mg twice daily for 12 weeks.
  Other Names: Metformin Group
  Arms: Metformin Group

SUMMARY:
This study is being done to compare the effect of regular exercise and metformin in people who have prediabetes. It is a community-based, open-label, randomized trial in which eligible participants will be divided into two groups. One group will do moderate physical exercise, and the other group will take metformin for 12 weeks. We will check their fasting blood sugar and HbA1c before and after the treatment to see which method works better for controlling sugar levels. The study is being done in a low-resource community setup to see which option is more practical and effective in real-life Pakistani settings.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 59 years
* Diagnosed with prediabetes based on ADA criteria (FPG: 100-125 mg/dL or HbA1c: 5.7-6.4%)
* Stable HbA1c levels (no significant fluctuation in the last 3 months)
* Body Mass Index (BMI) less than 30 kg/m²
* Willing and able to provide written informed consent
* Willing to participate in the assigned intervention (exercise or metformin) for 12 weeks
* Residing within the community and able to attend scheduled follow-ups

Exclusion Criteria:

* Age 60 years or older
* Diagnosis of Type 2 Diabetes Mellitus (T2DM) or use of anti-diabetic medications
* Family history of diabetes in first-degree relatives (parent or sibling)
* Known cardiovascular, renal, or hepatic disease
* Pregnancy or lactation
* Physical disability or limitation that would interfere with performing moderate-intensity exercise
* Uncontrolled hypertension (SBP ≥ 160 mmHg or DBP ≥ 100 mmHg)
* Known allergy or contraindication to metformin
* Alcohol or substance abuse

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 226 (Estimated)
Dates: Start 2025-08-10 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Change in Glycated Hemoglobin (HbA1c) from Baseline to 12 Weeks | Baseline and 12 week
  HbA1c (%) will be measured to assess glycemic improvement following 12 weeks of intervention.

SECONDARY OUTCOMES:
Weight change | Baseline to 12 weeks
  Change in weight in kilograms from baseline to 12 weeks following the two interventions

CONTACTS AND LOCATIONS:
Overall Officials: Umair Ali, Principal Investigator — CMH Nowshera
Locations (1):
- Department of Preventive Medicine, Combined Military Hospital Nowshera, Nowshera, Pakistan

IPD SHARING:
Plan to Share IPD: No
To maintain patients confidentiality